CLINICAL TRIAL: NCT04132128
Title: SUCCEED - Soroka Utility for Counting Carbs Easily and Effectively for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Idit Liberty MD, Head of Diabetes Clinic, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SOR- 0320-15 CTIL
Record Dates: First submitted 2019-08-07; First posted 2019-10-18 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Carbohydrates; Insulin Sensitivity; HbA1C
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: described in above section
Masking Description: no masking - open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- study (Experimental): 6 meetings with a dietician diabetes educator assimilating simple CC tool
  Interventions: Other: carbohydrate counting
- control (Other): meeting with dietician as needed with regular education of CC
  Interventions: Other: carbohydrate counting

INTERVENTIONS:
Other: carbohydrate counting — taught how to count carbohydrates in their diet with their personal tool

SUMMARY:
Counting Carbohydrates (CC) is the preferable method used to calculate the amount of insulin needed for a meal. This method is employed by patients with type 1 diabetes melitus (T1DM). the patients receive the general arithmetic calculation of how much insulin to inject for 15 grams/1 portion of carbohydrate (carb to insulin ratio (C:I) and insulin sensitivity (IS). However, Diabetes Educators are often confronted with difficulties guiding their T1DM patient when using this method and find patients get confused calculating the amount of carbs needed. The investigators sought to create a simple tool that would help our patients implement the CC method easily and properly.

DETAILED DESCRIPTION:
Objectives: To develop an easily understood CC tool accessible to all T1D patients.

Primary outcome - HbA1c at 3 and 6 months after intervention. Second primary - patients satisfaction with the tool.

Methods: The investigators created a tool which includes two tables with the patients' individual doses calculated by the clinics professional team, displaying his IS and C:I. The first table's values drive from the IS, showing how many insulin units should be given to correct blood sugar levels according to the measured result before the meal, and second drives from the patient's own C:I, which shows how many insulin units should be given according to the chosen food items. Blood glucose target is also decided on an individual basis. Together, with the patient, the investigators create a list containing only food items in one's personal diet with attached values. Protein dishes and fatty items such as oil or an egg appear with the value of zero insulin if that is the correct figure for the particular patient. After filling out the two tables, the investigators apply them in 8 steps 1-measure blood sugar, 2-find the right insulin correction dose according to the 1st table, 3-plan the meal, 4-find the insulin dose for the food items chosen, 5-combine the insulin dose of step 2+4, 6-injection insulin by pen or insulin pump, 7-consume the meal. 8-measure blood sugar 2 hours after meal to make sure the right dose was applied. At all visits the lists are discussed and missing food items are added. Using this tool enables to introduce CC to most patients.The tool has been applied in different languages: Hebrew, Arabic, Russian, English and Amharic and was used by patients whose individual learning skills varied over a very wide spectrum.

Patients were randomized into two groups. Group 1-received the new tool. Group 2-learned carb counting on customary basis. All participants met 6 times with a registered dietician diabetes educator to practice carb counting.

Data collected at recruitments and at the end of the study: HbA1c, daily insulin dosage, lipids profiles and questioners (PAID of WHO).

Subgroup analyses were done according to gender, diabetes years and education.

ELIGIBILITY:
Inclusion Criteria:

* men or woman with a clinical diagnosis of DM TYPE 1
* Age- >18
* Insulin treatment: pump or injection in basal- bolus system

Exclusion Criteria:

* No insulin treatment
* 8.5%> HbA1C.
* Pregnancy or Breastfeeding.
* Critical illness such as ens stage cancer or CHF
* Recurrent hospitalizations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months after intervention
  HbA1C for measuring glucose control

SECONDARY OUTCOMES:
patients satisfaction | 6 months after intervention
  patient questionnaire on satisfaction on quality of life. The scale is from 0 (no problem) to 4 (very problematic)
HbA1C for measuring glucose control | 3 months after intervention
  HbA1C for measuring glucose control

CONTACTS AND LOCATIONS:
Overall Officials: Shula Witko, Study Director — Diabetes Clinic Dietitian, Soroka University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Shula Vitko, Dietitian of Diabetes clinic
Supporting Information: Study Protocol